CLINICAL TRIAL: NCT03772444
Title: Use of Beetroot Juice to Protect Against Postoperative Ileus (POI) Following Colorectal Surgery: a Pilot Study.
Acronym: BEET IT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The pilot study was set up to assess whether the used dosing regimen of beetroot juice demonstrated to reach the therapeutic objective. The study was terminated early, as the deadline for the grant application for a larger study was approaching.
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EC/2017/1476
Record Dates: First submitted 2018-12-05; First posted 2018-12-11 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Postoperative Ileus
MeSH Terms: interventions — Water

STUDY DESIGN:
Masking Description: Patients undergoing colorectal surgery will be randomized (n=10) to receive one week daily 70 ml of beetroot juice (~ 7 mmol inorganic nitrate) or (n=10) an equivalent volume of nitrate-depleted beetroot juice (control group 1). An additional control group (n=10) is added to the pilot study, in which patients will receive an equivalent volume of water (control group 2); this allows us to investigate whether the antioxidants present in beetroot juice contribute to the protective effect of beetroot juice in POI. Beetroot juice and nitrate-depleted beetroot juice cause discoloration of urine (beeturia) and feces from the purple betacyanin pigments in beetroot; for the control group that receives water, this will not be the case and blinding for this group is thus not possible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Beetroot juice (Active Comparator)
  Interventions: Dietary Supplement: Beetroot juice
- Control group 1 (Placebo Comparator)
  Interventions: Dietary Supplement: Nitrate-depleted beetroot juice
- Control group 2 (Sham Comparator)
  Interventions: Dietary Supplement: Water

INTERVENTIONS:
Dietary Supplement: Beetroot juice — Patients will drink 70 ml of beetroot juice daily in the week prior to surgery; the last dose will be administered via the nasogastric tube just before the start of the procedure.
  Arms: Beetroot juice
Dietary Supplement: Nitrate-depleted beetroot juice — Patients will drink 70 ml of nitrate-depleted beetroot juice daily in the week prior to surgery; the last dose will be administered via the nasogastric tube just before the start of the procedure.
  Arms: Control group 1
Dietary Supplement: Water — Patients will drink 70 ml of water in the week prior to surgery; the last dose will be administered via the nasogastric tube just before the start of the procedure.
  Arms: Control group 2

SUMMARY:
The BEET IT study investigates the possible protective effect of beetroot juice on POI following colorectal surgery in (partially) blinded single-center phase 2 randomized trial (pilot study).

DETAILED DESCRIPTION:
Postoperative ileus (POI) is a transient impairment of gastrointestinal motility following abdominal surgery, which leads to increased morbidity, prolonged hospitalization and increased healthcare cost. The pathogenesis of POI involves inflammation and oxidative stress, similar to ischemia/reperfusion injury that can be counteracted with beetroot juice. Beetroot juice is a source of inorganic nitrate, which by conversion of nitrate to nitrite in the body, exerts its protective effect. We before demonstrated in a preclinical model that administration of exogenous nitrite was shown to protect against POI. The aim of this pilot study is to investigate the possible protective effect of beetroot juice ingestion on POI following colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

• All patients undergoing colonic or upper rectum laparoscopic surgery.

Exclusion Criteria:

* Pregnancy or breast feeding
* Psychiatric pathology capable of affecting comprehension and judgment faculty
* History of metastatic disease
* History of prior abdominal bowel surgery
* Abdominal radiation treatment
* Chronic constipation (defined as two or fewer bowel movements per week)
* Gut motility influencing agents (e.g. tricyclic antidepressants, chronic use of laxatives)
* Frequent use of mouthwash, as this affects the enterosalivary circulation of nitrate
* Current use of broad-spectrum antibiotics, which will affect the oral flora and likely affect the nitrate reductase activity
* More than one bowel anastomosis during this surgery

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-05-25 (Actual); Study Completion 2019-05-25 (Actual)

PRIMARY OUTCOMES:
Time until recovery of gastrointestinal function. | up to 30 days after surgery
  Recovery of gastrointestinal function is defined as the interval (in days) from the end of surgery until passage of stool AND tolerance of solid food.

SECONDARY OUTCOMES:
Time until passage of stool, flatus or until tolerance of (semi-)solid oral diet (in days). | up to 30 days after surgery
Overall post-operative complication rate defined according to the Clavien-Dindo Classification. | 3 months postoperatively
Presence of prolonged postoperative ileus. | up to 30 days after surgery
  Prolonged postoperative ileus is defined as presence of 2 or more of the following criteria on or after day 4 postoperatively: nausea or vomiting, inability to tolerate a solid or semi-solid oral diet, abdominal distension, absence of flatus and stool, radiological evidence of ileus.

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No